CLINICAL TRIAL: NCT00211653
Title: Single Center Randomized Clinical Trial of the Effects of Acetylcysteine in the Prevention of Postoperative Renal Failure
Brief Title: Acetylcysteine in the Prevention of Renal Failure After Bypass Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3212-B
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-09-19 (Estimated); Status verified 2007-09

CONDITIONS: Kidney Failure
Keywords: Kidney failure; Thoracic surgery; Acetylcysteine
MeSH Terms: conditions — Renal Insufficiency | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: N-Acetylcysteine

SUMMARY:
The purpose of this study is to determine if Acetylcysteine is effective in preventing renal failure associated with cardiac surgery

DETAILED DESCRIPTION:
Postoperative renal dysfunction is a predictor of significant morbidity and mortality among patients undergoing cardiac surgery. The mortality associated with coronary artery by-pass surgery increases from 2% to almost 19% in patients with renal failure and approaches 60% in patients who require hemodialysis. Patients with preoperative renal dysfunction referred for coronary artery by pass surgery have an extraordinarily high risk of requiring postoperative dialysis. For example, among those patients with preoperative creatinine >2.5 mg/dL, almost 50% require hemodialysis.

Comparison: N-Acetylcysteine is superior to placebo in preventing renal failure after cardiac surgery

ELIGIBILITY:
Inclusion Criteria:

* Pts with baseline chronic kidney disease (eGFR<60 ml/min/1.73m2)undergoing cardiac surgery

Exclusion Criteria:

* Patients on hemodialysis preoperatively
* IV contrast within 4 days prior to surgery
* Urgent/emergent surgery
* History of renal transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2003-04; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Rise in creatinine above baseline | 7 days postoperatively

SECONDARY OUTCOMES:
Creatinine increase >25% or =/> 0.5 mg/dl above baseline | Postoperative days 5, 7 and 30
Length of stay in the ICU and the hospital
Operative mortality | 30-day

CONTACTS AND LOCATIONS:
Overall Officials: Selcuk Adabag, MD, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Veterans Affairs Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Adabag AS, Ishani A, Koneswaran S, Johnson DJ, Kelly RF, Ward HB, McFalls EO, Bloomfield HE, Chandrashekhar Y. Utility of N-acetylcysteine to prevent acute kidney injury after cardiac surgery: a randomized controlled trial. Am Heart J. 2008 Jun;155(6):1143-9. doi: 10.1016/j.ahj.2008.01.013. Epub 2008 Mar 5. PMID 18513531